CLINICAL TRIAL: NCT03000829
Title: Code Blue Outcomes & Process Improvement Through Leadership Optimization Using Teleintensivists-Simulation
Acronym: COPILOT-Sim
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Intermountain Health Care, Inc. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: COPILOT-SIMULATION; 1050317 (Other: Intermountain Health IRB)
Record Dates: First submitted 2016-09-14; First posted 2016-12-22 (Estimated); Results first posted 2024-05-31 (Actual); Last update posted 2024-05-31 (Actual); Status verified 2023-12

CONDITIONS: Cardiac Arrest
Keywords: Code blue; Code team; Crisis team leadership; Cardiopulmonary resuscitation; Telemedicine; Simulation; Mock code; In-hospital cardiac arrest
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tele-intensivist consultation (Experimental): Standardized consultation to on-site cardiac arrest response team by off-site intensivist via two-way audiovisual link using a mobile telemedicine cart
  Interventions: Other: Tele-intensivist consultation
- Control (Placebo Comparator): Simulated "observation" by ICU physician by displaying a silent, pre-recorded, non-interactive videotape of an ICU physician. The on-site participants will be told that an intensive care physician is observing the mock code.
  Interventions: Other: Simulated "observation" by ICU physician

INTERVENTIONS:
Other: Tele-intensivist consultation — Standardized consultation to on-site cardiac arrest team by off-site intensivist via two-way audiovisual link using a mobile telemedicine cart
  Arms: Tele-intensivist consultation
Other: Simulated "observation" by ICU physician — Display of silent, pre-recorded, non-interactive videotape of an ICU physician. The on-site cardiac arrest team will be told that an intensive care physician is observing the mock code.
  Arms: Control

SUMMARY:
This multicenter randomized trial will employ in-situ cardiac arrest simulations ("mock codes") to test whether using telemedicine technology to add an intensive care physician as the "copilot" for cardiac arrest resuscitation teams influences chest compression quality, resuscitation protocol adherence, team function, and provider experience.

DETAILED DESCRIPTION:
Only 15-30% of patients who suffer in-hospital cardiac arrest (IHCA) survive to hospital discharge. Factors associated with lower mortality and improved function include provision of high-quality, minimally-interrupted chest compressions and swift defibrillation of eligible arrhythmias. Unfortunately, resuscitation teams provide suboptimal care to 25-40% of IHCA victims. A dedicated IHCA team "copilot" may improve resuscitation team performance by providing the team leader with parallel analysis, situational awareness augmentation, action checking, protocol verification, and error correction. Critical care physician involvement via a telemedicine link could allow experienced specialists to fill the "copilot" role in a cost and resource-efficient manner, particularly in smaller hospitals with fewer available physicians.

The current study will evaluate how consultation by an off-site intensive care physician via a telemedicine link influences local IHCA teams' quality of care, team function and provider experience during simulated cardiac arrest events ("mock codes").

ELIGIBILITY:
Inclusion criteria (on-site cardiac arrest team):

* Are 18 years of age or older

Inclusion criteria (teleintensivist cardiac arrest team copilot):

* Are 18 years of age or older
* Are a board-certified or board-eligible critical care physician
* Provide clinical care through the Intermountain Healthcare Telecritical Care program

Exclusion criteria (both groups):

* Are under 18 years of age
* Are a member of the study research team

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1001 (Actual)
Dates: Start 2016-12; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ithan Peltan, MD, Principal Investigator — Intermountain Health Care, Inc.
Locations (7):
- United States (7):
  - American Fork Hospital, American Fork, Utah
  - Intermountain Medical Center, Murray, Utah
  - The Orthopedic Specialty Hospital, Murray, Utah
  - McKay-Dee Hospital, Ogden, Utah
  - Park City Hospital, Park City, Utah
  - Riverton Hospital, Riverton, Utah
  - LDS Hospital, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be available, after relevant IRB approval, by application to the principal investigator and Intermountain Office of Research.

REFERENCES:
- [Background] Spielberger CD, Gorsuch RL, Lushene R, Vagg PR, Jacobs GA. Manual for the State-Trait Anxiety Inventory. Palo Alto, CA: Consulting Psychologists Press; 1983.
- [Background] Marteau TM, Bekker H. The development of a six-item short-form of the state scale of the Spielberger State-Trait Anxiety Inventory (STAI). Br J Clin Psychol. 1992 Sep;31(3):301-6. doi: 10.1111/j.2044-8260.1992.tb00997.x. PMID 1393159
- [Background] McKay A, Walker ST, Brett SJ, Vincent C, Sevdalis N. Team performance in resuscitation teams: comparison and critique of two recently developed scoring tools. Resuscitation. 2012 Dec;83(12):1478-83. doi: 10.1016/j.resuscitation.2012.04.015. Epub 2012 May 3. PMID 22561464
- [Background] Cooper S, Cant R, Porter J, Sellick K, Somers G, Kinsman L, Nestel D. Rating medical emergency teamwork performance: development of the Team Emergency Assessment Measure (TEAM). Resuscitation. 2010 Apr;81(4):446-52. doi: 10.1016/j.resuscitation.2009.11.027. Epub 2010 Feb 1. PMID 20117874
- [Result] Peltan ID, Guidry D, Brown K, Kumar N, Beninati W, Brown SM. Telemedical Intensivist Consultation During In-Hospital Cardiac Arrest Resuscitation: A Simulation-Based, Randomized Controlled Trial. Chest. 2022 Jul;162(1):111-119. doi: 10.1016/j.chest.2022.01.017. Epub 2022 Jan 19. PMID 35063451
- [Derived] Silva JAM, Mininel VA, Fernandes Agreli H, Peduzzi M, Harrison R, Xyrichis A. Collective leadership to improve professional practice, healthcare outcomes and staff well-being. Cochrane Database Syst Rev. 2022 Oct 10;10(10):CD013850. doi: 10.1002/14651858.CD013850.pub2. PMID 36214207

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: Simulation events
Groups:
- Tele-intensivist Consultation Cardiac Arrest Simulations: Standardized consultation to on-site cardiac arrest response team by off-site intensivist via two-way audiovisual link using a mobile telemedicine cart
  Tele-intensivist consultation: Standardized consultation to on-site cardiac arrest team by off-site intensivist via two-way audiovisual link using a mobile telemedicine cart
- Control Cardiac Arrest Simulations: Simulated "observation" by ICU physician by displaying a silent, pre-recorded, non-interactive videotape of an ICU physician. The on-site participants will be told that an intensive care physician is observing the mock code.
  Simulated "observation" by ICU physician: Display of silent, pre-recorded, non-interactive videotape of an ICU physician. The on-site cardiac arrest team will be told that an intensive care physician is observing the mock code.
- Telemedical Intensivist Consultants: Critical care physicians serving as consultants during simulation events randomized to tele-intensivist consultation
Period: Overall Study
Arm/Group | Tele-intensivist Consultation Cardiac Arrest Simulations | Control Cardiac Arrest Simulations | Telemedical Intensivist Consultants
Started | 521; 45 Simulation events | 466; 37 Simulation events | 14; 0 Simulation events
Completed | 521; 45 Simulation events | 466; 37 Simulation events | 14; 0 Simulation events
Not Completed | 0; 0 Simulation events | 0; 0 Simulation events | 0; 0 Simulation events

BASELINE CHARACTERISTICS:
Population: Unit of analysis is the "Simulation event." Demographic data was not collected for on-site simulation participants.
Units Other Than Participants: Simulation events
Groups:
- Total: Total of all reporting groups
Arm/Group | Tele-intensivist Consultation | Control | Total
Number analyzed (Participants) | 521 | 466 | 987
Number analyzed (Simulation events) | 45 | 37 | 82
Age, Customized [Count of Units; unit: Simulation events] — Population: Age of on-site simulation participants - not collected
  Simulation events
    Age | NA — Age not collected for individual simulation participants and not applicable to unit of analysis ("simulation events") | NA — Age not collected for individual simulation participants and not applicable to unit of analysis ("simulation events") | NA — Total not calculated because data are not available (NA) in one or more arms.
Sex: Female, Male [Count of Units; unit: Simulation events]
  Female | NA — Sex not collected for individual simulation participants and not applicable to unit of analysis ("simulation events") | NA — Sex not collected for individual simulation participants and not applicable to unit of analysis ("simulation events") | NA — Total not calculated because data are not available (NA) in one or more arms.
  Male | NA — Sex not collected for individual simulation participants and not applicable to unit of analysis ("simulation events") | NA — Sex not collected for individual simulation participants and not applicable to unit of analysis ("simulation events") | NA — Total not calculated because data are not available (NA) in one or more arms.
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
  Participants
    number analyzed (Participants) | 0 | 0 | 0
    (all) |  |  | 0
Region of Enrollment [Number; unit: participants]
  United States | 521 | 466 | 987

OUTCOME MEASURES:

1. Primary Outcome: Fraction of Pulseless Time With no Chest Compressions
Time Frame: From initiation of intervention or placebo control until completion of two complete cycles of CPR (an average of 4 minutes)
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available. Per protocol, simulations for which equipment malfunction precluded measurement of compression quality were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: Fraction analysis time CPR not delivered
Units Other Than Participants: simulation events
Arm/Group | Tele-intensivist Consultation | Control
Number analyzed (Participants) | 425 | 439
Number analyzed (simulation events) | 36 | 35
Fraction analysis time CPR not delivered | 0.22 (0.13) | 0.19 (0.10)
Statistical Analysis 1: Comparison: Tele-intensivist Consultation vs Control; Test type: Superiority; p = 0.41, t-test, 2 sided

2. Secondary Outcome: Time From Onset of Shockable Rhythm to Defibrillation
Time Frame: From onset of simulated VF or VT until first defibrillation or end of simulation
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available and resuscitation team delivered ≥1 shock to the mannequin during the simulation. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of protocol adherence were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Simulation events
Arm/Group | Tele-intensivist Consultation | Control
Number analyzed (Participants) | 353 | 394
Number analyzed (Simulation events) | 30 | 31
seconds | 37 (33) | 36 (25)
Statistical Analysis 1: Comparison: Tele-intensivist Consultation vs Control; Test type: Superiority; p = 0.86, t-test, 2 sided

3. Secondary Outcome: Fraction of Chest Compressions With Complete Release
Time Frame: as for outcome 1
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of compression quality were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: Fraction compression in analysis window
Units Other Than Participants: Simulation events
Arm/Group | Tele-intensivist Consultation | Control
Number analyzed (Participants) | 425 | 439
Number analyzed (Simulation events) | 36 | 35
Fraction compression in analysis window | 0.89 (0.14) | 0.89 (0.15)
Statistical Analysis 1: Comparison: Tele-intensivist Consultation vs Control; Test type: Superiority; p = 0.97, t-test, 2 sided

4. Secondary Outcome: Fraction of Chest Compressions at Target Rate
Time Frame: as for outcome 1
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Fraction compression in analysis window
Units Other Than Participants: Simulation events
Arm/Group | Control | Tele-intensivist Consultation
Number analyzed (Participants) | 439 | 425
Number analyzed (Simulation events) | 35 | 36
Fraction compression in analysis window | 0.59 (0.23) | 0.58 (0.29)
Statistical Analysis 1: Comparison: Control vs Tele-intensivist Consultation; Test type: Superiority; p = 0.87, t-test, 2 sided

5. Secondary Outcome: Time to First Dose of Epinephrine
Time Frame: From initiation of simulation through termination of simulation, an average of 15 minutes
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available and epinephrine was administered. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of protocol adherence were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: seconds
Units Other Than Participants: Simulation events
Arm/Group | Control | Tele-intensivist Consultation
Number analyzed (Participants) | 421 | 370
Number analyzed (Simulation events) | 33 | 31
seconds | 329 (130) | 344 (124)
Statistical Analysis 1: Comparison: Control vs Tele-intensivist Consultation; Test type: Superiority; p = 0.63, t-test, 2 sided

6. Secondary Outcome: Overall ACLS Protocol Adherence (Using Checklist Adapted From McEvoy ACLS Assessment Tool)
Time Frame: From initiation of simulation through termination of simulation, an average of 15 minutes
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of protocol adherence were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: Fraction of eligible actions performed
Units Other Than Participants: Simulation events
Arm/Group | Control | Tele-intensivist Consultation
Number analyzed (Participants) | 430 | 380
Number analyzed (Simulation events) | 34 | 32
Fraction of eligible actions performed | 0.77 (0.11) | 0.78 (0.12)
Statistical Analysis 1: Comparison: Control vs Tele-intensivist Consultation; Test type: Superiority; p = 0.62, t-test, 2 sided

7. Secondary Outcome: ACLS Protocol Errors (Using Checklist Adapted From McEvoy ACLS Assessment Tool)
Time Frame: From initiation of simulation through termination of simulation, an average of 15 minutes
Population: as for outcome 6
Measure: Mean (Standard Deviation); unit: Number of protocol errors
Units Other Than Participants: Simulation events
Arm/Group | Control | Tele-intensivist Consultation
Number analyzed (Participants) | 430 | 380
Number analyzed (Simulation events) | 34 | 32
Number of protocol errors | 2.8 (1.7) | 2.9 (1.4)
Statistical Analysis 1: Comparison: Control vs Tele-intensivist Consultation; Test type: Superiority; p = 0.84, t-test, 2 sided

8. Secondary Outcome: Team Emergency Assessment Measure Score
Description: The validated "Team Emergency Assessment Measure (TEAM)" evaluates non-technical performance of the on-site resuscitation team. The score (range 0-4) for each simulation was obtained by averaging the mean score for each of 11 component scores (each component item scored 0-4, with higher values representing better performance).
Time Frame: From initiation of simulation through termination of simulation, an average of 15 minutes
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of team performance were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: score on composite TEAM scale
Units Other Than Participants: Simulation events
Arm/Group | Control | Tele-intensivist Consultation
Number analyzed (Participants) | 421 | 370
Number analyzed (Simulation events) | 34 | 32
score on composite TEAM scale | 3.2 (0.6) | 3.3 (0.6)
Statistical Analysis 1: Comparison: Control vs Tele-intensivist Consultation; Test type: Superiority; p = 0.40, t-test, 2 sided

9. Secondary Outcome: Types of Input by Telemedical Intensivist Copilot
Time Frame: From initiation of simulation through termination of simulation, an average of 15 minutes
Population: Pre-specified analysis included completed simulations for which complete compression quality data were available. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of telemedical intensivist input were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Count of Units; unit: Simulation events
Units Other Than Participants: Simulation events
Arm/Group | Tele-intensivist Consultation
Number analyzed (Participants) | 380
Number analyzed (Simulation events) | 32
Simulation events
  Arrest etiology identification | 27
  Arrest etiology treatment | 24
  Medical record review | 26
  Role clarity for on-site team | 19
  CPR quality | 10

10. Secondary Outcome: Opinions of Study Subjects About Experience Participating in Simulated Cardiac Arrest, Using a Locally-developed and Validated Survey Instrument
Description: Measured domains: understanding of telemedicine intensivist copilot's role, beliefs about telemedicine intensivist copilot's ability to integrate with on site team, ability to influence on-site team performance, comfort with telemedicine intensivist copilot's role, and function of telemedicine interface
Time Frame: Immediately after simulation
Population: Pre-specified analysis included complete surveys returned by on-site participants in completed simulations for which complete compression quality data were available. Per protocol, simulations for which equipment malfunction or simulation error precluded measurement of resuscitation quality were excluded, as were intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Count of Participants; unit: Participants
Arm/Group | Tele-intensivist Consultation
Number analyzed (Participants) | 275
Participants
  Survey participant: "Telemedical intensivist consultation improved the resuscitation care quality." | 174
  Survey participant: "Telemedical intensivist consultation helped team function more smoothly." | 176

11. Secondary Outcome: Short-form State-Trait Anxiety Inventory Score
Description: The short-form State-Trait Anxiety Inventory (STAI) measures acute stress experienced by respondents using 6 questions (scores for each question range from 1 to 4, with higher values indicating more stress). Analyzed respondent-level values use the total score (range 4-24) obtained by summing the score for each of the six questions, with higher values indicating more respondent-reported acute stress.
Time Frame: Immediately after simulation
Population: Pre-specified analysis included completed surveys by participants completed simulations for which complete compression quality data were available. Per protocol, participants in simulations for which equipment malfunction or simulation error precluded measurement of compression quality were excluded, as were participants in intervention-group simulations classified as "run-in" simulations because they occurred before optimization of the telemedicine audio equipment.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Control | Tele-intensivist Consultation
Number analyzed (Participants) | 259 | 275
score on a scale | 12.9 (2.1) | 12.9 (1.9)
Statistical Analysis 1: Comparison: Control vs Tele-intensivist Consultation; Test type: Superiority; p = 0.92, Mixed Models Analysis

12. Secondary Outcome: Presence of Telemedicine Audiovisual Connection Problems for Intervention Group Simulation Event
Time Frame: From initiation of simulation through termination of simulation, an average of 15 minutes
Population: as for outcome 1
Measure: Count of Units; unit: Simulation events
Units Other Than Participants: Simulation events
Arm/Group | Tele-intensivist Consultation
Number analyzed (Participants) | 425
Number analyzed (Simulation events) | 36
Simulation events | 14

ADVERSE EVENTS:
Time Frame: Through completion of simulated cardiac arrest resuscitation and associated debriefing, an average of 30 minutes
Description: Study participants were medical personnel participating in simulated cardiac arrest resuscitation. All-cause mortality was not an applicable adverse event or outcome.
Arm/Group | Control | Tele-intensivist Consultation
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/466 | 0/521
Other Adverse Events (participants affected / at risk) | 0/466 | 0/521

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-07-10): https://cdn.clinicaltrials.gov/large-docs/29/NCT03000829/Prot_SAP_000.pdf